CLINICAL TRIAL: NCT06542666
Title: Cognitive Functional Therapy Versus Therapeutic Exercises for Treating Individuals With Chronic Shoulder Pain: A Pilot and Feasibility Study
Brief Title: Cognitive Functional Therapy for Chronic Shoulder Pain: Pilot and Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Danilo Harudy Kamonseki, Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 79422824.0.0000.5188
Record Dates: First submitted 2024-07-23; First posted 2024-08-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Shoulder Pain; Exercise Therapy; Psychosocial Rehabilitation
Keywords: Shoulder pain; Subacromial pain; Rotator cuff related pain; Shoulder Impingement; Chronic pain; Psychosocial; Rehabilitation; Biopsychosocial
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy (Experimental): Cognitive Functional Therapy will be conducted once a week, in individual and in-person sessions lasting approximately 40 minutes, over eight weeks.
  Interventions: Other: Cognitive Functional Therapy
- Exercises (Active Comparator): Twelve participants will be allocated to this group. They will perform strengthening and stretching exercises twice a week for eight weeks, with each session lasting approximately 30 to 40 minutes.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Cognitive Functional Therapy — The intervention focuses on addressing the maladaptive cognitive, physical, and lifestyle behaviors related to the disorder.
  Cognitive functional therapy will focus on factors considered to contribute to the pain disorder, addressing the following topics:
  1. The multidimensional nature of persistent pain, beliefs, emotions, and behaviors (movement and lifestyle) that can reinforce a vicious cycle of pain sensitization and disability.
  2. Specific functional training designed to normalize maladaptive and provocative postural and movement behaviors as directed by the individual's presentation.
  3. Targeted functional integration into daily activities that are avoided and/or provocative for the patient.
  4. Counseling on physical activity and lifestyle, which will include promoting a gradual increase in physical activity based on the individual's preference and availability, advice on sleep hygiene, stress management strategies, and social re-engagement
  Arms: Cognitive Functional Therapy
Other: Exercises — Individuals allocated to this group will perform stretching and strengthening exercises. The self-stretching exercises will target the upper trapezius and posterior shoulder region. Each stretching exercise will be performed for 3 repetitions of 30 seconds, with an interval of 10 seconds between repetitions.
  The strengthening exercises will be performed using resistance elastic bands. Three sets of 10 repetitions will be performed for each strengthening exercise, with 1 minute of rest between sets. The strengthening exercises will target the lower and middle trapezius, anterior serratus, and the external and internal rotators of the shoulder.
  Arms: Exercises

SUMMARY:
This pilot randomized controlled clinical trial (RCT) will assess the feasibility and identify the key components necessary for conducting the main RCT, which will involve the comparison of Cognitive Functional Therapy with Therapeutic Exercises in individuals with chronic shoulder pain. The main questions it aims to answer are:

* What barriers to the participation of the included individuals might arise?
* Will the assessment procedures and outcome measures be feasible and suitable?
* What time will be necessary to conduct the assessments?
* Will participants be willing to be randomized to the proposed treatment groups?
* What barriers to the clinical delivery of Cognitive Functional Therapy in the healthcare system might exist?
* Will the treatment(s) be acceptable to patients?
* Will participants adhere to the treatment?
* What will the recruitment rates be per week/month?
* Will there be any selection bias?
* Will participant retention be high among the allocation groups?
* Will the data be complete?
* What will the data variability be?
* Will the treatment effects/outcomes be consistent with expectations and previous literature?

DETAILED DESCRIPTION:
Shoulder pain is a potentially debilitating musculoskeletal condition, with functional, physical, and psychological impact. Its chronicity has been mainly correlated with affective-emotional and cognitive dimensions of pain. In this scenario, interventions for individuals with chronic shoulder pain should be seen within the biopsychosocial model. In this context, Cognitive Functional Therapy (CFT) emerges as a psychologically informed physiotherapeutic approach directed towards the biopsychosocial and multidimensional nature of pain, which is divided into three approaches to reduce pain and disability: (1) understanding pain, (2) controlled exposure, and (3) lifestyle change. The present study aims to verify the feasibility and viability of a randomized clinical trial to compare the effects of Cognitive Functional Therapy with therapeutic exercises in individuals with chronic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Age between 18 and 60 years;
* Presence of shoulder pain for more than 3 months;
* Pain intensity of 4 points or more on the 11-point Numeric Pain Rating Scale during the past week.
* High level of disability or moderate level of irritability.

Exclusion Criteria:

* History of fracture or surgery of the clavicle, scapula, and/or humerus, surgical stabilization or rotator cuff repair;
* History of dislocation, instability (positive sulcus sign or apprehension test), and/or rotator cuff tear (positive drop arm test);
* Adhesive capsulitis verified by the presence of gradual onset pain associated with stiffness and reduced passive and active mobility;
* Ongoing pregnancy;
* Reproduction of shoulder pain radiating to the entire upper limb during cervical or thoracic spine tests (positive Spurling test);
* Neurological or systemic diseases that may alter muscle strength and sensitivity such as rheumatoid arthritis, fibromyalgia, lupus, gout, and diabetes;
* Corticosteroid injection in the shoulder region in the last 3 months;
* Physiotherapy treatment in the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 8 weeks
  Analyze the ability to recruit 12 individuals per group, totaling a sample of 24 individuals with chronic shoulder pain;
Retention rate | 8 weeks
  This will be evaluated through individual follow-up by the responsible physiotherapist during the 8-week treatment period, during which the physiotherapist will fill out an attendance sheet at each session to also characterize the completion of the intervention by each participant;
Acceptability of the intervention | 8 weeks
  This will be estimated through adherence to the appointment schedule and mainly through questioning after each intervention session.

SECONDARY OUTCOMES:
Pain intensity | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  The pain will be measured with 11 point - Numerical Rating Pain Scale with scores ranging from 0 (no pain) to 10 (maximum pain).
Shoulder Pain and Disability Index | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  Shoulder disability will be measured with Shoulder Pain and Disability Index (SPADI), with score ranging from 0 to 100, with higher scores indicating greater shoulder disability.
Chronic Pain Self-Efficacy Scale | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  Self-efficacy will be measured using the Chronic Pain Self-Efficacy Scale (CPSS). The total score ranges from 30 to 300 points, with higher scores indicating greater self-efficacy.
Tampa Scale for Kinesiophobia | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  Kinesiophobia will be measured using the Tampa Scale for Kinesiophobia (TSK). The total score ranges from 17 to 68 points, with higher scores indicating worse beliefs about pain related to movement.
Pain Catastrophizing Scale | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  Pain catastrophizing will be measured using the Pain Catastrophizing Scale (PCS). The total score ranges from 0 to 52 points, with higher scores indicating greater pain catastrophizing.
Pittsburgh Sleep Quality Index | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 to 21 points. A score greater than 5 indicates poor sleep quality, with significant difficulty in at least two components of the questionnaire or moderate difficulty in three components.
Biopsychosocial aspects | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  Biopsychosocial aspects will be measured with short screening questions on biopsychosocial aspects of chronic pain.
Patients' expectations of the treatment. | Baseline
  For the assessment of patients' expectations regarding their treatment, participants will respond to the question, "How much do you expect your shoulder problem to change as a result of treatment?" Their responses will be measured on a 7-point Likert scale, where 1 corresponds to "worse" and 7 corresponds to "completely recovered."
Patient-Specific Functional Scale | Pre (baseline), 4 weeks, and post Treatment (8 weeks)
  The Patient-Specific Functional Scale (PSFS) will be used to assess functional status. Individuals will score on an 11-point scale, indicating how difficult it is to perform 3 to 5 activities that are important to them. A score of 0 on the 11-point scale indicates "unable to perform the activity," while a score of 10 indicates "able to perform the activity at the pre-injury level.

CONTACTS AND LOCATIONS:
Overall Officials: VALÉRIA MA OLIVEIRA, PhD, Principal Investigator — Universidade Federal da Paraíba
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared under request.

REFERENCES:
- [Derived] Gava V, da Silva Eugenio JM, Meziat-Filho N, Almeida LA, Maciel DG, do Nascimento JDS, de Andrade PR, Santos Fonseca RN, Medeiros Barbosa G, de Oliveira VMA, Kamonseki DH. Cognitive functional therapy versus therapeutic exercises for the treatment of individuals with chronic shoulder pain: A protocol for a randomized controlled trial. PLoS One. 2025 Apr 21;20(4):e0320025. doi: 10.1371/journal.pone.0320025. eCollection 2025. PMID 40258003